CLINICAL TRIAL: NCT05997719
Title: Exploring Cancer Evolution, Prognostic and Predictive Biomarkers in EGFR-mutant NSCLC
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, MD, Chief of Medical Oncology Department, Sun Yat-sen University
Other Study IDs: B2023-287-01
Record Dates: First submitted 2023-08-03; First posted 2023-08-18 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: EGFR mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue, blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate genomic architecture, cancer evolution and their relationship with clinical outcomes in EGFR-mutant NSCLC.

DETAILED DESCRIPTION:
EGFR mutations are detected in about 50% of East Asian NSCLC and 10% of Western NSCLC. EGFR-mutant NSCLC harbors distinct genomic architecture including high ITH, early diversification, genome instability, low background mutation rates. But despite its high ITH, EGFR-mutant NSCLC usually have better prognosis than NSCLC with other driver mutations even without the application of targeted therapies, indicating that EGFR mutations may have distinct impacts on cancer evolution. This study intends to investigate the genomic architecture, cancer evolution trajectories and their relationship with clinical outcomes in EGFR-mutant NSCLC, and to identify prognostic and predictive biomarkers for this population that could potentially guide therapeutic decisions and improved clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older
2. Histologically or cytologically confirmed non-small-cell lung cancer
3. ECOG PS=0-2
4. EGFR mutations confirmed by tissue or peripheral blood
5. Can provide tumor tissue samples (fresh or archived)
6. The subject should have good compliance, who would participate in the research voluntarily, and sign the informed consent

Exclusion Criteria:

1. History of other malignancies within 5 years (excluding basal cell carcinoma of the skin or other carcinoma in situ that has been resected).
2. Unable to provide sufficient tumor tissue for analysis.
3. Subjects with active, unstable systemic diseases, such as active infection, uncontrolled hypertension, heart failure (NYHA class >= II), unstable angina pectoris, acute coronary syndrome, severe arrythmia, severe liver, kidney or metabolic diseases, HIV infection.
4. Subjects who are deemed unable to comply with the study requirements or complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically or cytologically confirmed EGFR-mutant NSCLC
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Intratumor heterogeneity (ITH) | 5 years
  Intratumor heterogeneity in terms of genomic architecture, transcriptomic profiles and clonal composition; Investigate the relationship between ITH, clinical features and clinical outcomes in EGFR-mutant NSCLC

SECONDARY OUTCOMES:
Clinical utility of ctDNA in EGFR-mutant NSCLC | 5 years
  Clinical utility of ctDNA in dissecting ITH, and its relationship with clinical features and clinical outcomes in EGFR-mutant NSCLC

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guanzhou, China